CLINICAL TRIAL: NCT01131390
Title: What Ventilator Settings Are Most Comfortable for Patients With COPD or Obesity.
Brief Title: Ventilator Settings and Comfort
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bridgeport Hospital (Other)
Responsible Party: Constantine A. Manthous, MD, Bridgeport Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Bpthosp11001
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-03

CONDITIONS: Obesity; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Obesity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ventilator setting changes — Ventilator settings will be changed every 3 minutes as described above, simultaneously measuring respiratory mechanics and patients' comfort.

SUMMARY:
No studies have been done to examine whether patients with obstructive lung disease and obesity are more comfortable on some ventilator settings than on others. The purpose of the current study is to examine this question systematically.

DETAILED DESCRIPTION:
Methods: Demographic and physiologic data will be recorded. Investigators will begin measurements more than 60 minutes after last dose of sedative and measurements to occur when no major interventions are planned or medications are scheduled. Then patients will undergo the following ventilator settings (all of which are within ranges ordinarily employed) in random order for 3 minutes of each setting (pressures measured midway i.e. 1.5 minutes - at each interval to ensure safety; stopped if static airway pressure>30 cmH2O):

1. Assist control

   1. Tidal volumes of 6 ml/kg, 8 ml/kg and 10 ml/kg
   2. Flow regimes: constant (CF) and decelerating (dec) at 40, 60 and 80 L/min;
2. Pressure support (PS) 0, 10 and 20 cmH2O with PEEP=5 cmH2O

Patients will be randomized to receive the following in either forward or reverse order: CF60L/min in 6 then 8 then 10 ml/kg; then at 8 ml/kg CF40, Dec40, Dec60, CF60, CF80, Dec80; then PS=0, 10, 20 cmH2O.

In the last 30 second of each setting, patients will be asked to indicate their level of comfort (1-10 in increasing comfort) using a visual analog Borg Score (when they can see/write) or to indicate on their fingers when they cannot write.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 y) admitted to the MICU of Bridgeport Hospital on mechanical ventilation for:

  * Exacerbation of COPD (smoking history>20 pkyrs AND chest radiographic or function abnormalities supportive of the diagnosis); OR
  * Body mass index>40 kg/m2 and acute on chronic hypercapnic respiratory failure.
* Patients must be awake, not have received narcotics for more than 2 hours and possess capacity to consent themselves.
* Patients must have recovered sufficiently from their acute illness to be candidates for weaning per hospital protocol i.e. not in shock, no pressors and PaO2:FiO2>120.

Exclusion Criteria:

* Patients extubated for comfort care only.
* Patients with successful weaning trial that otherwise clinically requires extubation.
* Patients with unresolved pneumonia, unresolved congestive heart failure, neuromuscular disease or kyphoscoliosis-related respiratory failure will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Patients' comfort | 40 minutes
  Borg score of patients' dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Manthous, MD, Principal Investigator — Bridgeport Hospital
Locations (1):
- Bridgeport Hospital, Bridgeport, Connecticut, United States